CLINICAL TRIAL: NCT06876077
Title: Evaluation of the Effectiveness of Auricular Acupuncture in Improving Dry Eye Symptoms in University Students: A Randomized Controlled Trial
Brief Title: Evaluation of the Effectiveness of Auricular Acupuncture in Improving Dry Eye Symptoms in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Doctor of Philosophy, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2468/DHYD-HDDD
Record Dates: First submitted 2025-02-28; First posted 2025-03-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye Symptoms
Keywords: Auricular Acupuncture; Dry eye symptoms; University students
MeSH Terms: interventions — Acupuncture, Ear; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular acupuncture + Artificial Tears (Experimental): Auricular acupuncture is administered in each side of the ear for four weeks, with five sessions lasting five days each. Artificial tears were continuously administered over the four-week intervention period.
  Interventions: Other: Auricular acupuncture; Other: Artificial Tears (AT)
- Sham auricular acupuncture + Artificial Tears (Sham Comparator): Sham auricular acupuncture is administered in each side of the ear for four weeks, with five sessions lasting five days each. The artificial tear is continuously administered over the four-week intervention period.
  Interventions: Other: Sham auricular acupuncture; Other: Artificial Tears (AT)

INTERVENTIONS:
Other: Auricular acupuncture — Auricular acupuncture is administered in each side of the ear for 4 weeks using patches, each possessing a square shape with a side length of 10 mm, coupled with a sterilized needle measuring 0.25 x 1.3 mm. Five acupoints are selected on one ear, including the will be performed at Shenmen (TF4), Mu 1 (TG2b), Mu 2 (AT1b), Kidney (CO10), and Liver (CO12). These acupoints are believed to be effective in relieving dry eye symptoms. The patch will be kept on the auricle for 5 days and be replaced 5 times during the experimental period.
  Arms: Auricular acupuncture + Artificial Tears
Other: Sham auricular acupuncture — Sham auricular acupuncture is administered in each side of the ear for 4 weeks using patches, each possessing a square shape with a side length of 10 mm, without a needle. Five acupoints are selected on one ear, including the will be performed at Shenmen (TF4), Mu 1 (TG2b), Mu 2 (AT1b), Kidney (CO10), and Liver (CO12). These acupoints are believed to be effective in relieving dry eye symptoms. The patch will be kept on the auricle for 5 days and be replaced 5 times during the experimental period.
  Arms: Sham auricular acupuncture + Artificial Tears
Other: Artificial Tears (AT) — Artificial tear drops were applied 5-6 times per day over the 4-week period

SUMMARY:
Dry eye symptoms can cause various discomforts in the eyes and/or visual disturbances. This condition not only limits daily personal activities and reduces quality of life and mental health but also has negative economic impacts on families and society. Currently, complementary and alternative methods have been employed, with acupuncture being a promising treatment for patients with dry eye disease. Among these, auricular acupuncture has been proven effective in managing eye diseases and improving dry eye symptoms.

DETAILED DESCRIPTION:
Participants and Methods: A randomized controlled trial was conducted to evaluate the effectiveness of auricular acupuncture in improving dry eye symptoms by stimulating five acupoints: Auricular Shenmen (TF4), Eye 1 (TG2b), Eye 2 (AT1b), Liver (CO12), and Kidney (CO10), combined with the application of artificial tears 5-6 times per day for 4 weeks and the potential adverse effects of auricular acupuncture. A total of 50 participants were randomly assigned to 2 group (A and B) and the allocation ratio was 1:1. In group A: Participants received sham auricular acupuncture by sticking patches at specific points on one ear, combined with artificial tear drops. In group B: Participants underwent auricular acupuncture at the same points on one ear, combined with artificial tear drops. Stimulation was performed three times daily by pressing each needle or adhesive patch for approximately 10 seconds or until the ear turned red or became slightly painful. The total duration of the study was 4 weeks. Participants alternated auricular acupuncture or sham acupuncture between ears for five sessions, with each session lasting 5 days. Our study evaluate: (1) The improvement in dry eye symptoms acccording to the Ocular Surface Disease Index (OSDI) and the 5-item Dry Eye Questionnaire (DEQ-5); (2) The impact on quality of life was evaluated using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) and (3) Adverse effects during auricular acupuncture: Pain, allergy at the site of auricular acupuncture, acupuncture vertigo.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria:

* Be at least 18 years of age.
* Exhibit symptoms of dry eye, such as dryness, eye fatigue, eye itching, a foreign body sensation in the eye, burning or stinging sensations, blurry vision, light sensitivity, excessive tearing, or drooping eyelids.
* Have no refractive errors or related eye conditions.
* Visual acuity of both eyes ≥ 8/10 on the Snellen chart (normal vision).
* Show signs of dry eye with an OSDI score of ≥ 13 points
* Have never undergone auricular acupuncture before.
* Voluntarily agree to participate in the study.

Exclusion Criteria:

Participants must meet at least one of the following criteria:

* Have symptoms suggesting an acute infection or conditions affecting the conjunctiva, sclera, eyelids, cornea, or systemic diseases.
* Are using other methods to treat eye diseases.
* Have undergone eye-related surgery within the past 3 months.
* Have changed or worn contact lenses during the study period.
* Have inflamed or ulcerated skin in both ears.
* Are debilitated, exhausted, or have severe concomitant diseases.
* Are using medications affecting vision (diuretics, antihistamines, antihypertensives) or eye drops.
* Have a history of acupuncture vertigo.
* Are contraindicated with Sodium Hyaluronate.
* Are participating in other interventional studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Comparison of OSDI between auricular acupuncture at TF4, TG2b, AT1b, CO12 and CO10 points combined with artificial tear drops and Sham acupuncture at TF4, TG2b, AT1b, CO12 and CO10 points combined with artificial tear drops group | Baseline, Day 1, Day 6, Day 11, Day 16, Day 21 and Day 26
  The Ocular Surface Disease Index (OSDI) OSDI is a 12-item questionnaire that assesses dry eye symptoms occurring during the last week. The questions are divided into three sections which examine, respectively: subjective ocular symptoms, limitations in performing daily activities due to eye problems, and the influence of environmental conditions on eye comfort. Responses to every question ranged from 0, which represents "none of the time", to 4, which represents "all of the time". The final score ranges from 0 to 100 (sum of the 12 questions multiplied by 25 and divided by 12, and then rounded to the next integer) with higher scores representing greater disability: normal (0-12), mild (13-22), moderate (23-32), severe (33-100). A subject is classified as symptomatic when the total OSDI score is equal to or over thirteen points.

SECONDARY OUTCOMES:
Comparison of DEQ-5 between auricular acupuncture at TF4, TG2b, AT1b, CO12 and CO10 points combined with artificial tear drops and Sham acupuncture at TF4, TG2b, AT1b, CO12 and CO10 points combined with artificial tear drops group | Baseline, Day 1, Day 6, Day 11, Day 16, Day 21 and Day 26
  The 5-Item Dry Eye Questionnaire (DEQ-5) is a short subset of the full Dry Eye Questionnaire (DEQ) items which contains five questions regarding the frequency and intensity of eye discomfort, eye dryness and watery eyes in the past month. Responses are collected with two types of scales of the answers ranging from 0 to 4 or 5, with 0 corresponding to "never", and 4 with "constantly" in questions regarding the frequency of symptoms, or 0 with "never have it" and 5 with "very intense" in questions regarding the intensity of symptoms. The final score ranges from 0 to 22, a score > 6 suggests dry eye
Comparison of NEI VFQ-25 between auricular acupuncture at TF4, TG2b, AT1b, CO12 and CO10 points combined with artificial tear drops and Sham acupuncture at TF4, TG2b, AT1b, CO12 and CO10 points combined with artificial tear drops group | Baseline, Day 1, Day 6, Day 11, Day 16, Day 21 and Day 26
  The National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25) is composed of 25 items designed to assess visual disability and health-related quality of life. It contains 12 subcategories: general health, general vision, ocular pain, near vision activities, distance activities, social functioning, mental health, role difficulties, dependency, driving, color vision and peripheral vision. The questionnaire has a total score ranging from 0 to 100 (a higher score indicates better vision-specific quality of life).

OTHER OUTCOMES:
Adverse effects during auricular acupuncture | During procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Center HCMC - Branch no.3, Ho Chi Minh City, Ho Chi Minh, Vietnam

REFERENCES:
- [Background] Wrobel-Dudzinska D, Osial N, Stepien PW, Gorecka A, Zarnowski T. Prevalence of Dry Eye Symptoms and Associated Risk Factors among University Students in Poland. Int J Environ Res Public Health. 2023 Jan 11;20(2):1313. doi: 10.3390/ijerph20021313. PMID 36674068
- [Background] Hou PW, Hsu HC, Lin YW, Tang NY, Cheng CY, Hsieh CL. The History, Mechanism, and Clinical Application of Auricular Therapy in Traditional Chinese Medicine. Evid Based Complement Alternat Med. 2015;2015:495684. doi: 10.1155/2015/495684. Epub 2015 Dec 28. PMID 26823672
- [Background] Tan JY, Molassiotis A, Wang T, Suen LK. Adverse events of auricular therapy: a systematic review. Evid Based Complement Alternat Med. 2014;2014:506758. doi: 10.1155/2014/506758. Epub 2014 Nov 10. PMID 25435890
- [Background] Zhang CS, Yang AW, Zhang AL, May BH, Xue CC. Sham control methods used in ear-acupuncture/ear-acupressure randomized controlled trials: a systematic review. J Altern Complement Med. 2014 Mar;20(3):147-61. doi: 10.1089/acm.2013.0238. Epub 2013 Oct 19. PMID 24138333
- [Background] Huang Q, Zhan M, Hu Z. Auricular Acupressure for Dry Eye Disease: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Medicina (Kaunas). 2023 Jan 16;59(1):177. doi: 10.3390/medicina59010177. PMID 36676806
- [Background] Asiedu K, Kyei S, Boampong F, Ocansey S. Symptomatic Dry Eye and Its Associated Factors: A Study of University Undergraduate Students in Ghana. Eye Contact Lens. 2017 Jul;43(4):262-266. doi: 10.1097/ICL.0000000000000256. PMID 26963438
- See also: The Effects of Auriculotherapy on Relieving Symptoms of Dry Eye Syndrome — http://www.jkssh.or.kr/journal/view.html?doi=10.15434/kssh.2018.31.3.178